CLINICAL TRIAL: NCT02607917
Title: Testing a Community Intervention to Increase Aspirin Use for Primary Prevention of Cardiovascular Disease
Brief Title: Testing a Community Intervention to Increase Aspirin Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1201M8921
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Myocardial Infarction; Stroke
Keywords: Cardiovascular Disease
MeSH Terms: conditions — Myocardial Infarction; Stroke; Cardiovascular Diseases | interventions — Culture Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mass Media plus clinic intervention. (Experimental): These geographic areas will receive the media plus clinic intervention over a two year period.
  Interventions: Other: Mass Media plus clinic intervention.
- Media (Experimental): These geographic areas will receive the media intervention over a two year period.
  Interventions: Other: Media
- No Intervention (No Intervention): Adjacent states will receive no intervention.

INTERVENTIONS:
Other: Mass Media plus clinic intervention.
  Arms: Mass Media plus clinic intervention.
Other: Media
  Arms: Media

SUMMARY:
This research will test the effect of mass media or mass media plus a clinic based education program will improve appropriate aspirin use for cardiovascular disease prevention. It is a group randomized design of 24 geographic areas in Minnesota with adjacent states serving as controls.

DETAILED DESCRIPTION:
Proposed is a demonstration and implementation project to increase the appropriate use of aspirin for primary prevention of acute myocardial infarction and stroke in the population of Minnesota. Although significant progress in the reduction of acute myocardial infarction and stroke is apparent, these cardiovascular disorders continue as the leading causes of morbidity and mortality. In recent years, and in the context of the positive results from large randomized clinical trials, there is growing consensus that aspirin, when appropriately used, reduces cardiovascular morbidity in men aged 45-79 and women aged 55-79 years. The use of aspirin for primary prevention was recommended in the U.S. Preventive Services Task Force Report in 2009 and more recently in the CDC/CMS 'Million Hearts' ABCs (aspirin, blood pressure, cholesterol, smoking) campaign. Aspirin use is also recommended in the Healthy People 2020 goals. However, many adults who would benefit, are not taking aspirin.

The investigators have been fortunate to receive a large philanthropic donation to launch a campaign to increase appropriate aspirin use in the State of Minnesota. The proposed grant requests funding to evaluate that campaign and the innovative approaches it proposes. In the context of a innovative mass media effort, the investigators intend to test new methods for health system change to increase appropriate aspirin use. Using a two-arm design, the investigators have defined 24 geographic areas in the state that will form the basis for a group-randomized trial. This design will allow us to distinguish the effects of the intervention methods. The interventions will be evaluated by sequential surveys of the target-age general population at baseline and follow-up. Appropriate aspirin use in that population will be the primary goal and endpoint. Simultaneous surveys of adjacent Upper Midwestern states (Iowa, North and South Dakota, Wisconsin) will assess secular trends. Morbidity and mortality data will monitor disease trends and complications associated with aspirin use.

A substantial pilot study in a middle sized community in Northern Minnesota allows us to refine and validate our intervention and measurement methods at the community level. This pilot also demonstrated behavior change of a magnitude supportive of our design assumptions.

This program, if successful, should result in a generalizable program tested in a real world population setting.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men age 45-79.
* Healthy women age 55-79
* per USPSTF 2009 recommendations

Exclusion Criteria:

* History of cardiovascular disease
* aspirin allergy
* serious life-limiting illness

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10800 (Actual)
Dates: Start 2015-02-16 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Appropriate aspirin use. | 4-5 years
  Aspirin use will be determined by standardized surveys of randomly selected adults.

SECONDARY OUTCOMES:
Cardiovascular disease morbidity | 4-5 years
  Collected from hospital records of the Minnesota Hospital Association.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Roeser S, Duval S, Luepker RV, Eder M, Finnegan JR, Van't Hof JR. Population cessation of aspirin use for the prevention of cardiovascular disease. Am J Prev Cardiol. 2025 Feb 8;21:100941. doi: 10.1016/j.ajpc.2025.100941. eCollection 2025 Mar. PMID 40103687
- [Derived] Luepker RV, Eder M, Finnegan JR, Van't Hof JR, Oldenburg N, Duval S. Association of a Community Population and Clinic Education Intervention Program With Guideline-Based Aspirin Use for Primary Prevention of Cardiovascular Disease: A Nonrandomized Controlled Trial. JAMA Netw Open. 2022 May 2;5(5):e2211107. doi: 10.1001/jamanetworkopen.2022.11107. PMID 35536579
- [Derived] Duval S, Van't Hof JR, Oldenburg NC, Eder M, Finnegan JR Jr, Luepker RV. A community-based group randomized trial to increase aspirin use for primary prevention of cardiovascular disease: Study protocol and baseline results for the "Ask About Aspirin" initiative. Contemp Clin Trials Commun. 2021 Apr 19;22:100772. doi: 10.1016/j.conctc.2021.100772. eCollection 2021 Jun. PMID 34027223
- [Derived] Krzyzanowski B, Manson SM, Eder MM, Kne L, Oldenburg N, Peterson K, Hirsch AT, Luepker RV, Duval S. Use of a Geographic Information System to create treatment groups for group-randomized community trials: The Minnesota Heart Health Program. Trials. 2019 Mar 28;20(1):185. doi: 10.1186/s13063-019-3284-9. PMID 30922358